CLINICAL TRIAL: NCT00969449
Title: An Open Label, Randomized, Two-Way Crossover Trial to Compare the Pharmacokinetic Parameters of an Extended- Release Naproxen Sodium Tablet Relative to Naprelan® Tablets Following Single Dose Administration Under Fasted Conditions
Brief Title: Pharmacokinetics Study Comparing Naproxen Sodium Extended Release and Naprelan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14566
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Pharmacokinetics
Keywords: Naproxen Sodium
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Naproxen Sodium, (BAY H6689)
- Arm 2 (Active Comparator)
  Interventions: Drug: Naprelan, (BAY H6689)

INTERVENTIONS:
Drug: Naproxen Sodium, (BAY H6689) — One dose of Naproxen sodium extended release 660 mg under fasting conditions
  Arms: Arm 1
Drug: Naprelan, (BAY H6689) — One dose of Naprelan 500 mg (2 tablets) under fasting conditions
  Arms: Arm 2

SUMMARY:
To compare the pharmacokinetic profile of the proposed extended- release tablet of naproxen sodium 660 mg relative to two tablets of Naprelan 500 mg following single dose administration for 36 hours under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 55 years of age inclusive with a Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera®, or a double barrier and have a negative pregnancy test at Screening and Day 0 for each Dosing Period. Female subjects of non-childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Be willing to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the clinical protocol

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), naproxen sodium, or acetaminophen, and similar pharmacological agents or components of the products
* Females who are pregnant or lactating
* Loss of blood in excess of 500 ml within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury)
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases or malignancies
* Positive alcohol or drug test at Screening and on Day 0 of each Dosing Period
* Have taken any medications (except acceptable forms of birth control) within 10 days prior to dosing or throughout the trial, unless in the opinion of the Investigator and the Sponsor, the medication will not interfere with the trial procedures, data integrity, or compromise the safety of the subject
* Have taken ASA, ASA-containing products, acetaminophen (acetyl-para-amino-phenol or APAP) or any NSAID (OTC or prescription) 7 days prior to dosing or during the treatment period, other than trial treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of Naproxen Sodium ER 660 mg compared to Naprelan | 36 hours

SECONDARY OUTCOMES:
To assess safety and tolerability of the extended release naproxen sodium | 36 hours
To assess additional pharmacokinetic parameters | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States